CLINICAL TRIAL: NCT04381975
Title: Move in Mind: Program for Reducing Musculoskeletal Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Key collaborator, who would have delivered the intervention, moved abroad
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Barbel Knauper, James McGill Professor of Psychology, McGill University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Musculoskeletal Pain; Chronic Pain
MeSH Terms: conditions — Musculoskeletal Pain; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Move in Mind Program (Experimental): The Move in Mind Program is a 6-week Rolfing®-based intervention program shortened from ten to six sessions and adapted to a group setting by Rolfing® instructor Monica Canducci.
  Interventions: Behavioral: Move in Mind Program
- 6 Week Waitlist Control (Other): Participants will be crossed over to the Move in Mind program following the 6-week waitlist control. Participants of the waitlist control group will be asked to complete follow-up questionnaires both at the same time as the intervention group (after week six) as well as after their own program.
  Interventions: Behavioral: 6 Week Waitlist Control

INTERVENTIONS:
Behavioral: Move in Mind Program — Each of the six Move in Mind sessions will take place once a week for approximately 1.5 hours, with 12-17 individuals participating per class. The material and exercises taught will include physical floor exercises, breathing exercises, as well as awareness training.
  Arms: Move in Mind Program
Behavioral: 6 Week Waitlist Control — The waitlist control group will receive the Move in Mind program after 6 weeks.
  Arms: 6 Week Waitlist Control

SUMMARY:
The present pilot study will explore the range of mental and physical health benefits associated with a Rolfing®-based intervention program ("Move in Mind"). To assess the effects of this program on pain management and various psychological outcomes, the investigator's study will be offered to individuals with mild chronic musculoskeletal pain (e.g., lower back pain, neck pain, shoulder pain, knee pain, arthritic pain). Shortened from ten to six sessions and adapted to a group setting by Rolfing® instructor Monica Canducci, the intervention will be delivered weekly by Ms. Canducci, who is certified in Rolfing®. The program will target the potential associations of the Move in Mind program with better pain management (primary outcome) as well as increased body awareness and presence, increased well-being, and better stress management (secondary outcomes). Interested participants will be asked to complete a battery of questionnaires and psychometric scales to assess the variables of interest before (baseline) and after their participation in the Move in Mind program (six-week follow-up). A waitlist control group will also be assessed at baseline and follow-up and will then receive the Move in Mind sessions subsequently and also assessed after their participation.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* experiencing a type of mild musculoskeletal pain (e.g., pain related to the muscles, ligaments, bones, joints, or nerve compression)

Exclusion Criteria:

* pregnant
* receiving treatment for severe chronic pain
* have had recent concussions or fractures as a result of accidents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in quality and intensity of pain at the end of treatment/waitlist period. | 7 days after last intervention session in week six
  The short-form McGill Pain Questionaire (SF-MPQ) is a 15-item self-report measure that assesses the quality and intensity of a patient's pain. Descriptors either represent the sensory dimension (items 1-11; e.g., "Stabbing") or the affective dimension of pain experience (items 12-15; e.g., "Punishing-Cruel"). Patients respond to the SF-MPQ using an intensity scale ranging from 0 (none) to 3 (severe).

SECONDARY OUTCOMES:
Difference in changes in physical and mental health at the end of treatment/waitlist period. | 7 days after last intervention session in week six
  12-item Short Form Health Survey (SF-12 version)
Difference in perceived stress at the end of treatment/waitlist period. | 7 days after last intervention session in week six
  The Perceived Stress Scale is a 10-item scale measuring the degree to which situations in the past month are perceived as overwhelming or unpredictable.
Difference in positive and negative affect at the end of treatment/waitlist period. | 7 days after last intervention session in week six
  The Positive and Negative Affect Schedule (PANAS)
Difference in depressive disorder diagnoses and depressive symptom severity at the end of treatment/waitlist period. | 7 days after last intervention session in week six
  Patient Health Questionnaire (PHQ-9)
Difference in satisfaction with Move in Mind program at the end of treatment/waitlist period. | 7 days after last intervention session in week six
  8 items based on Frayn et al. (2020). Items such as "The program was easy to follow" or "I can see myself using what I learned in the program in the long term" are rated on a 5-point Likert-type scale from 1 (strongly disagree) to 5 (strongly agree).